CLINICAL TRIAL: NCT06757283
Title: Evaluation of Typhoid Conjugate Vaccine (TCV) Effectiveness Among Bangladeshi Children Using the Test-negative Design
Brief Title: ZyVac-TCV Bangladesh Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-24059
Record Dates: First submitted 2024-12-20; First posted 2025-01-03 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Typhoid Vaccination; Typhoid; Typhoid Fever
Keywords: Conjugate vaccine; Immunogenicity; Safety; Typhoid fever; Bangladesh; Children
MeSH Terms: conditions — Typhoid Fever | interventions — Carrier Proteins

STUDY DESIGN:
Intervention Model Description: This will be a phase III effectiveness study of the typhoid conjugate vaccine (Vi-TCV) (ZyVac® TCV). The study will be conducted in a closed cohort population of children aged 6 months to 15 years residing in a selected geographical catchment area in Dhaka, Bangladesh using a test-negative design (TND).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culture-positive case (Experimental): Eligible febrile patients who will be positive by blood culture for Salmonella enterica serotype Typhi and symptoms developed >14 days after vaccination, or, if unvaccinated, >14 days after the midpoint of the vaccination period.
  Interventions: Biological: Purified Vi capsular polysaccharide of Salmonella typhi conjugated to tetanus toxoid as carrier protein (Typhoid Vi Conjugate Vaccine I.P.). Trade name: ZyVac® TCV
- Culture-negative control (Active Comparator): Eligible febrile patients who will be negative by blood culture for Salmonella enterica serotype Typhi and symptoms developed >14 days after vaccination, or, if unvaccinated, >14 days after the midpoint of the vaccination period.
  Interventions: Biological: Purified Vi capsular polysaccharide of Salmonella typhi conjugated to tetanus toxoid as carrier protein (Typhoid Vi Conjugate Vaccine I.P.). Trade name: ZyVac® TCV

INTERVENTIONS:
Biological: Purified Vi capsular polysaccharide of Salmonella typhi conjugated to tetanus toxoid as carrier protein (Typhoid Vi Conjugate Vaccine I.P.). Trade name: ZyVac® TCV — Purified Vi capsular polysaccharide of Salmonella typhi conjugated to tetanus toxoid as carrier protein (Typhoid Vi Conjugate Vaccine I.P.)

SUMMARY:
This is a prospective closed cohort, open-label, phase III effectiveness study using a test-negative design of a typhoid conjugate vaccine, ZyVac® TCV (purified Vi capsular polysaccharide of Salmonella Typhi conjugated to tetanus toxoid as carrier protein), manufactured by Zydus Lifesciences Limited. The study will be conducted in a closed cohort population among children aged 6 months to 15 years residing in wards 5, 6, 7, 48, 49, 50, 63, 71, and 72 of Dhaka South City Corporation (DSCC). The targeted number of age-eligible children in the study area is ~92,000 among them ~60,000 will be vaccinated. A subset of the first 600 consenting participants will be selected by age strata (6 months to <2 years, 2-4 years, 5-15 years) for enrollment in the immunogenicity study with an additional three follow-up visits. Diary cards will be used to collect adverse events (AEs) following immunization (AEFI) data up to day 7 for a subset of active follow-up of the first 600 vaccinated participants. Participants not in this subset will be encouraged to go to the 'Adverse Event Monitoring Cell' at the Maniknagar field office. Data on serious adverse events (SAEs) will be reported for six months after vaccination. All study updates including AEs and SAEs will be reported to the data safety and monitoring board (DSMB) and sponsor. Passive surveillance for typhoid fever will be carried out in the Maniknagar field office and Mugda Medical College and Hospital in the catchment area among the age-eligible children.

DETAILED DESCRIPTION:
This will be a phase III effectiveness study of the typhoid conjugate vaccine (Vi-TCV) (ZyVac® TCV). The study will be conducted in a closed cohort population of children aged 6 months to 15 years residing in a selected geographical catchment area in Dhaka, Bangladesh using a test-negative design (TND). The TND is a particular type of case-control study including controls who present themselves with similar signs and symptoms (to those of the cases) in the same healthcare facilities. Individuals with the disease of interest are tested with a laboratory assay where test-positive and test-negative individuals are considered cases and controls, respectively.

Hypothesis:

The typhoid Vi-polysaccharide conjugate vaccine will be effective in preventing typhoid fever among Bangladeshi children.

Specific Objectives

Primary objective:

To evaluate the effectiveness of typhoid conjugate vaccine (TCV) against blood culture-confirmed typhoid fever using the test-negative design

Secondary objective:

To evaluate the effectiveness of typhoid conjugate vaccine (TCV) against blood culture-confirmed typhoid fever stratified by age groups (6 months to <2 years, 2 to 4 years, 5 to 15 years) To evaluate the effectiveness of typhoid conjugate vaccine (TCV) against blood culture-confirmed typhoid fever stratified by the period of follow-up (first and second six months) after vaccination To determine the immunogenicity of TCV in a subset of participants, stratified by age groups (6 months to <2 years, 2 to 4 years, 5 to 15 years)

Study area The study will be conducted in wards 5, 6, 7, 48, 49, 50, 63, 71, and 72 of Dhaka South City Corporation, covering an area of ~10.33 km2. No TCV campaigns have been conducted in this area. According to the Population and Housing Census 2022, the total population within the selected geographical catchment area is ~465,000 with households of ~122,000. The proportion of males is 54 percent and the average household size is ~3.8 people. Assuming ~20% of the population is from the 6-month to 15-year age group, the expected number of age-eligible children is ~92,000.

Baseline mapping A map of the study area will be created based on open-source georeferenced satellite images (source: Esri, Maxar, Earthstar Geographics, and the geographical information system (GIS) user community). The satellite image of the study area will be printed by separating it into several small pieces and provided to the field team for data collection. In this process field team will visit the entire area according to the map and draw the structure/building, road, and other salient geographic features in the printed images. A unique geographical information system (GIS) identification number will be assigned for all the buildings/structures, and submitted to the GIS team to develop the digital vector data (point, line, and polygon feature). The digital data of structure/building (polygon feature) centroid x and y coordinates will be used to represent real-world coordinate values or global positioning system (GPS) values.

Baseline listing All households in the study area will be assigned a unique identification number and all household members will be enumerated. Information about the age-eligible children including name, age, sex, date of birth, and parent's name will be obtained. In addition, the name of the HH head, address, and cell phone number of HHs will be collected. The previously assigned GIS ID will be incorporated into the baseline listing form and the newly identified structure will be updated in the GIS database. We will take photos of birth certificates or national immunization cards to confirm the age of participants if available. Verbal consent will be provided by either the head of the household or a key informant.

Participant card for potentially eligible children for vaccination After preparing the baseline list, we will identify the age-eligible (6 months to 15 years) participants. Then we will prepare participant cards for all eligible children which will be provided before the vaccination. There will be a unique identification number on the participant card which will be used during vaccination. A master list of potential eligible participants will be prepared.

Vaccination

Temporary exclusion criteria for vaccination:

Participants will be temporarily excluded from being vaccinated if, at the point of vaccination, any of the following apply:

Receipt of any other vaccines in the last 30 days Current temperature of at least 38oC or reported fever within 24 hours prior to vaccination Use of antipyretics within 4 hours prior to vaccination Unmarried girls between the ages of ≥12 to 15 years old whose first day of their last menstrual period (LMP) is more than 28 days ago or who do not know the date they last menstruated upon presentation

If these apply, the participant will be temporarily excluded from vaccination until the temporary exclusion criteria no longer apply. Please note, for children with fever above 38oC this must be a minimum of 48 hours after the fever has resolved. Unmarried girls between the ages of ≥12 to 15 years whose first day of their LMP is more than 28 days or who do not know the date they last menstruated upon presentation will be asked to return after starting their next menstruation for vaccination. A re-assessment will be conducted to ensure these temporary exclusion criteria no longer exist.

Verification of the potentially eligible children All the households that have age-eligible children will be informed to visit the nearest vaccination centre. If a participant's birth certificate or national immunization cards were not provided during the baseline listing, we will notify their parents or guardians to bring them during vaccination. After arrival at the vaccination centre, the participant and vaccination ID will be verified with the listing database and the master list. Then the screening will be carried out according to inclusion/exclusion criteria.

Informed consent The latest approved version of written informed consent/assent will be presented to the participant's parent/guardian in the local language detailing no less than the exact nature of the study, what it will involve for the participant, the implications and constraints of the protocol, the known side effects and any risks involved in taking part. It will be clearly stated that the participant's parent/guardian is free to withdraw their child from the study at any time for any reason without prejudice to future care, without affecting their legal rights, and with no obligation to give the reason for withdrawal. The participant and their parents/guardians will be allowed as much time as they wish to consider the information, within the recruitment period, and the opportunity to question the investigator or other independent parties to decide whether they will participate in the study. Written informed consent/assent will then be obtained, with additional opt-in consent for blood specimen, using participants' parent/guardian's dated signature or thumbprint and dated signature of the person who presented and obtained the informed consent. Information sheets will be given to children aged 11 -15 years in a language that they can understand. The person obtaining consent will record informed assent on the consent form, for children aged 11 and older. The person who obtained the consent must be suitably qualified and experienced and have been authorized to do so by the Principal Investigator (PI). A copy of the signed informed consent will be given to the participant. The original signed form will be retained at the study site. A third party will act as a witness for the parent/guardian to attest that the information in the consent form and any other written information was accurately explained to, and understood by the parent/guardian and that informed consent was freely given by the parent/guardian. The witness will also sign and date the consent form.

Screening and eligibility assessment An informed written consent will be obtained after confirming the participants by checking the database. After proper consenting process, a temperature will be taken and parents will be asked about antipyretic use and timings of previous vaccination to assess temporary exclusion criteria. A brief medical history will be taken and eligibility will be assessed against inclusion and exclusion criteria. Participants with temporary exclusion criteria will be informed and asked to return 48 hours after the fever has resolved or 30 days after the last vaccination was given for repeat assessment and re-consent. Unmarried girls between the ages of ≥12 to 15 years whose first day of their LMP is more than 28 days or who do not know the date they last menstruated upon presentation will be asked to return after starting their next menstruation, for vaccination. A member of the study team will collect/edit demographic information (including age and address) and participant contact details by screening case report form (CRF). After completion of the eligibility checking, a sticker will be allocated for the participant which includes the information of vaccination ID and temperature; these will be used in the vaccine accountability log.

Vaccination The vaccination team will finally check the identification and then administer the vaccine. After vaccination, information will be recorded in the vaccination CRF. If the participant is included in the immunogenicity study, a blood sample will be taken by a suitably trained staff member before vaccination. After administration of the study vaccine, participants will be asked to wait at least 30 minutes for any immediate hypersensitivity reactions or any other adverse events (AEs). The female participants of reproductive age should have been advised not to be pregnant within three months after the vaccination.

Investigational Medicinal Product (IMP) Purified Vi capsular polysaccharide of Salmonella typhi conjugated to tetanus toxoid as carrier protein (Typhoid Vi Conjugate Vaccine I.P.). Trade name: ZyVac® TCV, Zydus Lifesciences Limited.

Each 0.5ml vaccine dose contains:

Purified Vi-capsular polysaccharide of S.typhi 25 μg Conjugated to tetanus toxoid (carrier protein) 16 to 50 μg 2-Phenoxyethanol (as preservative) 2.50 mg Isotonic buffer solution q.s. The vaccine is packaged as a pre-filled 2.5ml 5-dose vial. It will be administered as an intramuscular injection preferably in the anterolateral aspect of the middle thigh for younger children, or the upper arm for older children with aseptic precautions.

Supply The Vi-TCV vaccine (ZyVac® TCV) will be provided by Zydus Lifesciences Limited.

Storage The Vi-TCV study vaccine will be stored at 2º to 8º C in a temperature monitored icddr,b cold room facilities, when not in use for daily activities. The vaccines will be stored in temperature-monitored refrigerators or cool boxes, when in use for daily activities. Each vial will be labeled with a "vaccine vial monitor"(VVM); a temperature-sensitive dot that provides an indication of the cumulative heat to which the vial has been exposed. It warns the end-user when exposure to heat is likely to have degraded the vaccine beyond an acceptable level and should not be used.

Special precautions for storage Store at 2°C to 8°C. Do not freeze. Discard if frozen. Keep out of reach of children. Shake gently before use. Do not use the vaccine after the expiration date shown on the label

Accountability of the study vaccine The vaccines will be shipped to a central storage facility in Bangladesh and passed through customs. It will then be transported and distributed to local vaccination sites whilst maintaining the cold chain (aiming for a temperature between 2º-8ºC). The number of doses of study vaccines that are received, used, and wasted will be documented daily during the study and checked weekly.

Adverse events following immunization After administration of the study vaccine, participants will be observed closely for at least 30 minutes for any immediate hypersensitivity reactions or any other adverse events (AEs). All details will be recorded in the CRF.

Adverse events follow up (Day 7, -1/+7):

A subset of 600 participants will be selected for active surveillance follow-up and the immunogenicity sub-study. A diary card will be given to each participant on the day of vaccination. Participants will be contacted by telephone or in-person after seven days of vaccination for follow-up and to record any adverse events following immunization (AEFI). The selection of these participants will be age-stratified (6 months to <2 years, 2-4 years, and 5-15 years) with an allocation of 200 in each age stratum.

Parents of participants not in this subset will be encouraged to go to the 'adverse event monitoring cell' at the Maniknagar field office which will have a medical doctor and also available on-call 24 hours a day for adverse event monitoring throughout the whole vaccination period + 7 days.

Information will include:

Verbal reconfirmation of consent for participation in the study. Report from parent/guardian of adverse events related to vaccination and use of medications following vaccination.

After administration of TCV, solicited local AEs (pain, redness, swelling and induration) and solicited systemic AEs (fever, nausea, vomiting, diarrhea, headache1, malaise1, myalgia1, arthralgia1, abnormal crying2, loss of appetite2, drowsiness2 and irritability2 (1: applicable for subjects aged ≥2 years; 2: applicable for subjects <2 years of age)) will be recorded for 7 days after vaccination.

Unsolicited (other) AEs will be recorded for 28 days after vaccination. Reiteration of contact details and instructions to attend the Maniknagar field office in case of fever (≥2 days and/or temperature

* 38°C at presentation).

Causality

The relationship of each adverse event to the study medication must be determined by a medically qualified individual according to the following definitions:

Related: There is suspicion that there is a relationship between the study vaccine and the AE (without determining the extent of probability); there is a reasonable possibility that the study vaccine contributed to the AE

Not related: There is no suspicion that there is a relationship between the study vaccine and the AE; there are other more likely causes and administration of the study vaccine is not suspected to have contributed to the AE Procedures for recording adverse events

From vaccination through day 7 After administration of TCV, solicited local AEs (pain, redness, swelling and induration), solicited systemic AEs (fever, nausea, vomiting, diarrhea, headache1, malaise1, myalgia1, arthralgia1, abnormal crying2, loss of appetite2, drowsiness2 and irritability2 (1: applicable for participants aged ≥2 years; 2: applicable for participants <2 years of age)) for 7 days after vaccination. Unsolicited (other) AEs will be recorded for 28 days after vaccination.

For injectable vaccines, the local signs and symptoms to be documented usually include, as a minimum, pain, redness, and swelling at the injection site in all age groups. Measuring devices of various types may be used to record the extent of redness and swelling. Fever will be documented using digital thermometers and axillary temperature will be determined. For subjective symptoms (for example, fatigue and myalgia) following scoring system will be considered.

All adverse events related to vaccination, as judged by a medically qualified investigator, occurring during the first 7 days post-vaccination that are observed by the study team/investigator or reported by the participant's parent/guardian, will be recorded on the CRF. The information will be collected both passively and actively.

For active surveillance of a subset of 600 participants, information will be actively collected via phone calls or home visits. Parents of participants not in this subset will be encouraged to go to the 'Adverse Event Monitoring Cell' at the Maniknagar field office which will have a medical doctor and also available on-call 24 hours a day for adverse event monitoring throughout the whole vaccination period + 7 days.

The following information will be recorded: description, date of onset and end date, severity, assessment of relatedness to study medication, and action taken. Follow-up information should be provided as necessary.

The severity of events will be assessed on the following scale: 1 = mild, 2 = moderate, 3 = severe, 4 = Potentially life-threatening

All Serious Adverse Events (SAEs) observed by the Investigators, members of the study team, or reported by the parent/guardian will be recorded on CRFs.

Throughout the study period Serious Adverse Events (SAEs), as judged by a medically qualified investigator, observed by the investigator, or members of the study team, or reported by the parent/guardian, will be recorded on the CRF. The following information will be recorded: description, date of onset and end date, severity, assessment of relatedness to study medication, and action taken. Follow-up information should be provided as necessary. All SAEs will be recorded in the CRFs, for the entire study duration. Participants with SAEs will be followed by a medically qualified investigator either until resolution or the event is considered stable.

Reporting procedures for serious adverse events The forms developed by the icddr,b institutional review board (IRB) will be used for reporting all SAEs.

All SAEs occurring within the 6 months post-vaccine administration will be reported to the Data Safety Monitoring Board (DSMB), Directorate General of Drug Administration (DGDA), the PI, and the other study investigators within 24 hours of the site study team becoming aware of the event. A more detailed report form will be completed and sent within the shortest period of the initial report, to all parties mentioned above. Additional and further requested information (follow-up or corrections to the original case) will be detailed in subsequent safety report forms. All SAEs must be reported to the study sponsor within 7 days. Summary reports will be submitted to the icddr,b IRB, and DGDA at the end of the study.

Indication for antipyretics and analgesics Antipyretics will be used in case of fever (axillary temperature >38◦C/100.4◦F or feels hot to touch) following vaccination. Analgesics will be used in case of pain, or discomfort after getting vaccinated.

Safety monitoring committee A DSMB will also be formed to oversee the safety component of the study. The DSMB members will not be involved in the study in any way. In addition, a physician with relevant study-related or therapeutic expertise will be identified as an independent safety monitor (ISM). The ISM will not be an investigator for this study. Under any circumstances, the identified ISM would be requested to carry out an independent assessment of the child presented with adverse events. The assessment details will be reported to the PI and DSMB.

Pregnancy follow-up Follow-up on pregnancy outcomes will be conducted for all married girls identified during routine follow-up as either being pregnant at the time of vaccination or becoming pregnant within three months of vaccination. This follow-up will include monthly visits until the end of the pregnancy, with the final contact occurring after delivery or pregnancy outcome. Starting from the eighth month of gestation, additional weekly follow-ups will be conducted via phone calls. We will record pregnancy-related information considering it as a medically important event.

Immunogenicity study A subset of 600 participants will be enrolled in the immunogenicity sub-study and will have an additional three face-to-face follow-up visits at the field office at one month (D30/+7 days), at 6 months (D180+/-14 days), and at one year (D365+/-30 days) after vaccination. The first 200 participants from each age stratum (6 months to <2 years, 2 to 4 years, 5 to 15 years) who give their consent will be selected and enrolled for the immunogenicity sub-study.

At these additional visits, the following procedures will be performed:

Confirmation of continued participation in the study Collection of blood (3ml for 6 months to 4 years and 5ml for 5 to 15 years ) Confirmation of contact details and reiteration of instructions to attend the health care facilities in case of fever for ≥2 days and/or temperature ≥38°C at presentation.

The above information will be recorded in the immunogenicity CRF. Parents/guardians of participants enrolled in the immunogenicity study will be given details of the follow-up appointments.

Surveillance for enteric fever Surveillance for enteric fever will be undertaken at the Maniknagar field office and Mugda Medical College and Hospital for all age-eligible (from 6 months to 15 years) residents recorded in the baseline list. Participants with a subjective history of ≥2 days of fever and/or a temperature of ≥38°C at presentation will be enrolled in the surveillance. A blood sample (3ml) will be collected for microbiological culture. The participants will receive appropriate clinical management. Blood culture-positive patients will be visited at home to confirm their identity, and collect information about their illness and patients will be asked to visit the field office if their condition is not improved. The treatment will be adjusted as necessary, based on laboratory testing.

Study staff will visit households, included in the baseline listing, periodically, to remind them to seek treatment at the Maniknagar field office if their children (both vaccinees and non-vaccinees) develop a fever.

Eligibility criteria for enrollment in the passive surveillance

Participants information, available in the listing database Parent/guardian is willing and competent to provide informed consent. For participants aged 11 to 15 years, informed assent will also be considered Participants from the study area who experienced a fever lasting for ≥2 days and/or temperature ≥38°C at presentation Participants aged 6 months to 15 years on the first day of the vaccination campaign

Laboratory procedures

Passive surveillance samples Microbiological culturing of blood samples collected from enrolled participants will be carried out using BACTEC or BacT/ALERT systems in the icddr,b Clinical Microbiology, Immunology and Molecular Diagnostic Laboratory. The sensitivity and specificity of the blood culture method are 59% and 100% respectively. Organisms from the suspected colonies will be identified by the biochemical tests and final identification will be done by slide agglutination test with Salmonella-specific antisera (Denka Sieken, Tokyo, Japan). The pattern of antibiotic susceptibility of Salmonella Typhi and Salmonella Paratyphi causing enteric fever will be assessed by the disk diffusion method on a Mueller-Hinton agar plate with Oxoid disks containing ampicillin, cotrimoxazole, chloramphenicol, azithromycin, ceftriaxone, ciprofloxacin, nalidixic acid, and cefixime. The procedure will be carried out following GCP guidelines and standard operating procedures. The results of these tests will be recorded in the participant CRF. The isolated strain will be preserved at the Mucosal Immunology and Vaccinology Laboratory for further analysis.

Immunogenicity study samples Blood samples taken for the immunogenicity sub-study will be transported to the icddr,b laboratory daily. The samples will be processed and stored by trained study staff, following standard operating procedures (SOP). The serum/plasma will be stored and used to measure the anti-Vi-IgG antibody using a commercially available Enzyme-linked Immunosorbent Assay (ELISA) kit (VaccZyme, The Binding Site). This assay will be performed according to the manufacturer's instructions. Laboratory processes will be conducted at the Mucosal Immunology and Vaccinology Laboratory at the icddr,b.

Withdrawal of participants Participants' parents/guardians can withdraw consent at any point. The investigator may also discontinue a participant from the study at any time if the investigator considers it necessary for any reason including: Ineligibility (either arising during the study or retrospectively having been overlooked at screening) Significant protocol deviation Significant non-compliance with treatment regimen or study requirements An adverse event or disease progression resulting in the inability to continue to comply with study procedures and follow-up

Depending on which aspects participants wish to withdraw from, the withdrawal will result in the cessation of any follow-up calls, visits, or blood tests (as applicable to the subset). No further treatment is required in the study, so no additional action will need to take place. Participants' parents/guardians will have the choice when withdrawing, to withdraw from active study procedures only (follow-up calls and visits) but remain in passive surveillance for the primary outcome, (allowing us to access their hospital records and blood test results), or withdraw from all study contact. Data and blood samples collected prior to the time of participant withdrawal will be kept and analyzed as part of the study data. A participant who withdraws from the study has the option to re-engage at a future date if they choose to do so. All participants who withdraw from the study will be given information on how to re-engage with the study if they so choose. Reasons for withdrawal from the study, if known, will be recorded in the participant's CRF.

Source documentation Each participant will have a complete source documentation of records including CRF, lab reports, and test results for the entire study period.

Data management The investigators will populate the content of participants' CRFs and all the study data will be recorded directly into an Electronic Data Capture (EDC) system (e.g. Octalsoft). Electronic devices and hard copies of CRFs will be used to collect and record data. Data will be collected online and uploaded to a cloud server regularly when electronic devices are brought back to the central field office, and reliable internet is available. Paper CRFs (pCRFs) will also be available as backup, in case of interruption of online data collection, pCRFs will be used for collecting data and data will then be entered into the EDC system when feasible.

Baseline listing data will be collected offline on an electronic device with an internally designed Android application database SQLite and SQL Server. The system will have some logical checks incorporated in the system and it will be checked before saving to the server. Data will be checked periodically using the SQL scripts for detecting errors. Errors will be corrected by the user and transferred to the server again. An audit trail of correction will always be available in the system after correction of data. Data management staff will keep backups from the SQL server database regularly and store the backup on the desktop, laptop, and other removable devices.

All other CRFs will be designed and maintained on EDC system, named Octalsoft, a secure web application for building and managing online surveys and databases. Quality control checks of the system will be performed on a regular basis. Both the EDC system (CRF data) and internally designed Android application will use a relational database via a secure web interface with data checks applied during data entry to ensure data quality.

All participants will be identified by a unique trial-specific number of and/or codes; this will not include any identifiable information. Some personal information will be saved on the Android application designed by icddr,b. Only site research staff and sponsor data managers will have access to view the personal information.

Trial staff will have access to both the internally designed Android application and Octalsoft via a unique username and password. Each trial staff member will have an appropriate level of access to CRFs and collected data, according to their roles and responsibilities within the trial.

All participant data will be stored and maintained on local servers in icddr,b as mentioned above for the duration of the trial. Anonymized data will be shared with the sponsor in India. At the end of the trial, all individually identifiable data will be removed, and fully anonymized data will be retained for further analysis.

Sample Size Calculation and Outcome A sample size of 515 (103 cases and 412 controls) will be required in this case-control test-negative design study assuming vaccine effectiveness of 80%, vaccine coverage of 65% in the target age-eligible population (6 months to 15 years), 4 controls per case, precision width of ± 10% (20%) and type 1 error rate of 0.05. Considering the incidence rate for typhoid fever of 230 per 100,000 person-years among the non-vaccinated population aged 6 months to 15 years, the target number of vaccinations is ~60,000.

To achieve the target number of vaccinees aged 6 months to 15 years representing ~31% of the total population), the required age-eligible children and population of all age groups will be ~92,000 and ~297,000 respectively.

Statistical analysis For the evaluation of vaccine protection, a conditional logistic regression model will be used, considering matched case-control status as the outcome and vaccination status and selected covariates as independent variables, taking non-receipt of vaccine as the referent category for assessment of vaccine protection. Odds ratios for the associations between vaccination and typhoid fever will be estimated by exponentiation of the coefficient for vaccination from the fitted model, and the standard error of the coefficient will be used to calculate 95% confidence intervals for the estimated effect. Protective effectiveness will be calculated as [(1 - odds ratio) X 100%]. The threshold of statistical significance will be considered at P <0.05.

Analysis of immunogenicity and safety data Geometric Mean Titres (GMT) and seroconversion rate (≥4-fold rise of anti-Vi-IgG antibody titre induced on day 30 compared to day 0 before vaccination) of anti-Vi-IgG antibody titre will be calculated. Analysis of covariance will be used to adjust for imbalances in baseline titres.

ELIGIBILITY:
Inclusion Criteria:

* Participant was included in the baseline list of the study population
* Participants living within the study catchment area at the time of vaccination
* Parent/guardian is willing and competent to provide informed consent (if the participant is 11 to 15 years of age, assent will also be sought)
* Participants aged between 6 months to15 years (i.e. up to 15 years 364 days) at the time of vaccination
* Apparently healthy (no complaints of febrile illness) on the day of vaccination
* Parent/guardian confirms that their child will be willing and be able to comply with study requirements

Exclusion Criteria:

* Has knowingly received a typhoid vaccine in the past
* Known allergy to any vaccine in the past
* Medical or social reasons that will prevent the participant from conforming to the study requirements as judged by a medical professional
* Planning to move away from the catchment area within the next 12 months
* Pregnant at the time of vaccination, as confirmed by a urine test (urine pregnancy test will be done in girls who are married)
* Confirmed or suspected immunosuppressive or immunodeficiency disorder; or subjects on any immunosuppressive or immunostimulant therapy
* Subject participated in another clinical study in the past 3 months

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 12 months
  Blood culture-confirmed typhoid fever

SECONDARY OUTCOMES:
Secondary outcome | 12 months
  Anti-Vi-IgG antibody concentration Blood culture-confirmed paratyphoid fever
Secondary outcome | 12 months
  Blood culture-confirmed paratyphoid fever

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The global burden of typhoid fever — https://pubmed.ncbi.nlm.nih.gov/15298225/
- See also: The global burden of typhoid and paratyphoid fevers: a systematic analysis for the Global Burden of Disease Study 2017 — https://pubmed.ncbi.nlm.nih.gov/30792131/
- See also: Antillón, M., et al., The burden of typhoid fever in low- and middle-income countries: A meta-regression approach. — https://pubmed.ncbi.nlm.nih.gov/28241011/
- See also: Meiring, J.E., et al., Burden of enteric fever at three urban sites in Africa and Asia: a multicentre population-based study. — https://pubmed.ncbi.nlm.nih.gov/34798028/
- See also: Ochiai, R.L., et al., A study of typhoid fever in five Asian countries: disease burden and implications for controls. — https://pubmed.ncbi.nlm.nih.gov/18438514/
- See also: World Health, O., Typhoid vaccines: WHO position paper, March 2018 - Recommendations. — https://pubmed.ncbi.nlm.nih.gov/29661581/
- See also: Qamar, F.N., et al., Adverse events following immunization with typhoid conjugate vaccine in an outbreak setting in Hyderabad, Pakistan. — https://pubmed.ncbi.nlm.nih.gov/32201138/
- See also: TyVAC. Currently available typhoid vaccines. 2023 — https://www.coalitionagainsttyphoid.org/the-issues/typhoid-vaccines/
- See also: GAVI. Typhoid conjugate vaccine (TCV) support. [cited 2024 14 April] — https://www.gavi.org/types-support/vaccine-support/typhoid
- See also: Typhoid vaccines: WHO position paper. — https://pubmed.ncbi.nlm.nih.gov/18260212/
- See also: Mond, J.J., A. Lees, and C.M. Snapper, T cell-independent antigens type 2. — https://pubmed.ncbi.nlm.nih.gov/7612238/
- See also: Weintraub, A., Immunology of bacterial polysaccharide antigens. — https://pubmed.ncbi.nlm.nih.gov/14670715/
- See also: Acharya, I.L., et al., Prevention of typhoid fever in Nepal with the Vi capsular polysaccharide of Salmonella typhi. — https://pubmed.ncbi.nlm.nih.gov/3657877/
- See also: Klugman, K.P., et al., Protective activity of Vi capsular polysaccharide vaccine against typhoid fever. — https://pubmed.ncbi.nlm.nih.gov/2890805/
- See also: Yang, H.H., et al., Efficacy trial of Vi polysaccharide vaccine against typhoid fever in south-western China. — https://pubmed.ncbi.nlm.nih.gov/11477965/
- See also: Froeschle, J.E. and M.D. Decker, Duration of Vi antibodies in participants vaccinated with Typhim Vi (Typhoid Vi polysaccharide vaccine) in an area not endemic for typhoid fever. — https://pubmed.ncbi.nlm.nih.gov/20003920/
- See also: Michel, R., et al., Outbreak of typhoid fever in vaccinated members of the French Armed Forces in the Ivory Coast. — https://pubmed.ncbi.nlm.nih.gov/16119438/
- See also: Pasetti, M.F., et al., Immunology of gut mucosal vaccines. — https://pubmed.ncbi.nlm.nih.gov/21198669/
- See also: Cryz, S.J., Jr., et al., Safety and immunogenicity of Salmonella typhi Ty21a vaccine in young Thai children. — https://pubmed.ncbi.nlm.nih.gov/8432597/
- See also: Simanjuntak, C.H., et al., Oral immunisation against typhoid fever in Indonesia with Ty21a vaccine. — https://pubmed.ncbi.nlm.nih.gov/1681365/
- See also: Levine, M.M., et al., Large-scale field trial of Ty21a live oral typhoid vaccine in enteric-coated capsule formulation. — https://pubmed.ncbi.nlm.nih.gov/2883393/
- See also: Olanratmanee, T., et al., Safety and immunogenicity of Salmonella typhi Ty21a liquid formulation vaccine in 4- to 6-year-old Thai children. — https://pubmed.ncbi.nlm.nih.gov/1634818/
- See also: Szu, S.C., et al., Laboratory and preliminary clinical characterization of Vi capsular polysaccharide-protein conjugate vaccines. — https://pubmed.ncbi.nlm.nih.gov/7927707/
- See also: Lin, F.Y., et al., The efficacy of a Salmonella typhi Vi conjugate vaccine in two-to-five-year-old children. — https://pubmed.ncbi.nlm.nih.gov/11320385/
- See also: Thiem, V.D., et al., The Vi conjugate typhoid vaccine is safe, elicits protective levels of IgG anti-Vi, and is compatible with routine infant vaccines. — https://pubmed.ncbi.nlm.nih.gov/21411598/
- See also: Safety and immunogenicity of a Vi polysaccharide-tetanus toxoid conjugate vaccine (Typbar-TCV) in healthy infants, children, and adults in typhoid endemic areas: a multicenter, 2-cohort, open-label, double-blind, randomized controlled phase 3 study — https://pubmed.ncbi.nlm.nih.gov/25870324/
- See also: WHO. Schistosomiasis. — https://www.who.int/news-room/fact-sheets/detail/schistosomiasis
- See also: WHO. Weekly Epidemiological Record. 2017; 2:13-20. 2007 — http://www.who.int/wer
- See also: Safety and Efficacy of a Typhoid Conjugate Vaccine in Malawian Children. — https://pubmed.ncbi.nlm.nih.gov/34525285/
- See also: Qadri, F., et al., Protection by vaccination of children against typhoid fever with a Vi-tetanus toxoid conjugate vaccine in urban Bangladesh: a cluster-randomised trial. — https://pubmed.ncbi.nlm.nih.gov/34384540/
- See also: Theiss-Nyland, K., et al., Assessing the Impact of a Vi-polysaccharide Conjugate Vaccine in Preventing Typhoid Infections Among Nepalese Children: A Protocol for a Phase III, Randomized Control Trial. — https://pubmed.ncbi.nlm.nih.gov/30845329/
- See also: WHO. INFORMATION SHEET OBSERVED RATE OF VACCINE REACTIONS TYPHOID VACCINE — https://cdn.who.int/media/docs/default-source/pvg/global-vaccine-safety/typhoid-vaccine-rates-information-sheet.pdf?sfvrsn=706de51b_4&download=true
- See also: Ng'eno, E., et al., Dynamic Incidence of Typhoid Fever over a 10-Year Period (2010-2019) in Kibera, an Urban Informal Settlement in Nairobi, Kenya. — https://pubmed.ncbi.nlm.nih.gov/37253442/
- See also: ASTMH — https://www.ajtmh.org/configurable/content/journals$002ftpmd$002f109$002f1$002farticle-p22.xml?t:ac=journals%24002ftpmd%24002f109%24002f1%24002farticle-p22.xml
- See also: Limited, Z.L. Summary of Product Characteristics as per Annexure C Typhoid vi Conjugate Vaccine I.P. ZyVac® TCV. — https://zyduslife.com/research
- See also: Antillon, M., et al., The Relationship Between Blood Sample Volume and Diagnostic Sensitivity of Blood Culture for Typhoid and Paratyphoid Fever: A Systematic Review and Meta-Analysis. — https://pubmed.ncbi.nlm.nih.gov/30307563/
- See also: Islam, M.T., et al., Use of Typhoid Vi-Polysaccharide Vaccine as a Vaccine Probe to Delineate Clinical Criteria for Typhoid Fever. Am J Trop Med Hyg, 2020. 103(2): p. 665-671 — https://pubmed.ncbi.nlm.nih.gov/32588803/

DOCUMENTS (1):
  • Study Protocol (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT06757283/Prot_000.pdf